CLINICAL TRIAL: NCT03257709
Title: The Arthroscopic Labral Excision or Repair Trial (ALERT) - A Randomised Controlled Trial to Determine the Effectiveness of Arthroscopic Hip Labral Surgery
Brief Title: The Arthroscopic Labral Excision or Repair Trial (ALERT)
Acronym: ALERT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Oxford (Other)
Collaborators: Arthritis Research UK (Other); The Royal College of Surgeons of England (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRAS 184490
Record Dates: First submitted 2017-01-04; First posted 2017-08-22 (Actual); Last update posted 2017-08-22 (Actual); Status verified 2017-08

CONDITIONS: Acetabular Labrum Tear

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arthroscopic acetabular labral repair (Active Comparator): Acetabular labral tear will be identified and reattached using suture anchors until a stable repair is achieved. If evidence of FAI is present ie: a cam or pincer lesion is identified then this will be treated with osteochondroplasty (cam) or acetabular rim recession (pincer).
  Interventions: Procedure: Arthroscopic acetabular labral repair
- Arthroscopic acetabular labral resection (Active Comparator): The acetabular labral tear will be identified and its' limits defined. The torn portion of labrum will be resected to a stable edge. As with arm 1 there will be treatment of FAI if identified.
  Interventions: Procedure: Arthroscopic acetabular labral resection

INTERVENTIONS:
Procedure: Arthroscopic acetabular labral repair — Acetabular labral tear will be identified and reattached using suture anchors until a stable repair is achieved. If evidence of FAI is present ie: a cam or pincer lesion is identified then this will be treated with osteochondroplasty (cam) or acetabular rim recession (pincer).
  Other Names: Labral Repair; Labral Reconstruction
  Arms: Arthroscopic acetabular labral repair
Procedure: Arthroscopic acetabular labral resection — The acetabular labral tear will be identified and its' limits defined. The torn portion of labrum will be resected to a stable edge. As with arm 1 there will be treatment of FAI if identified.
  Other Names: Labral Resection; Labral Debridement
  Arms: Arthroscopic acetabular labral resection

SUMMARY:
This study compares two established surgical treatments for acetabular labral tears. Patients will be prospectively recruited and randomised to either labral repair or debridement. All patients will be followed for 2 years after intervention with a primary outcome assessment at 6 months.

DETAILED DESCRIPTION:
STUDY DESIGN

Study design This will be a two-arm randomised controlled parallel group superiority study and will take place in a hospital setting. Stratification will be performed for sex and age by means of a minimisation technique during randomisation for each subject entering the trial.

Study population:

Adults between 18 and 75 years of age diagnosed with symptomatic acetabular labral tears demonstrated on MRI arthrogram but without radiographic evidence of OA ie: Kellgren & Lawrence grade less than 2 randomly selected from the Nuffield Orthopaedic Centre outpatient clinics.

Arm 1 Arthroscopic acetabular labral repair.

Arm 2 Arthroscopic acetabular labral resection

48 patients per arm (total 96 patients) will be selected from outpatient clinics and the operative waiting list (pre-operative assessment clinics) at the Nuffield Orthopaedic Centre, Oxford. The surgeries will be conducted using routine instrumentation in use at the centre.

STUDY PROCEDURES

Recruitment

All patients will undergo surgery in accordance with established practice regardless of their treatment allocation. Arthroscopy will be performed using standard anterior and lateral portals for insertion of instruments. All patients will undergo arthroscopic evaluation of the entire joint. Subsequent procedures will vary according to treatment allocation:

* Arm 1 - Labral Repair - acetabular labral tear will be identified and reattached using suture anchors until a stable repair is achieved. If evidence of FAI is present ie: a cam or pincer lesion is identified then this will be treated with osteochondroplasty (cam) or acetabular rim recession (pincer).
* Arm 2 - Labral Resection - the acetabular labral tear will be identified and its' limits defined. The torn portion of labrum will be resected to a stable edge. As with arm 1 there will be treatment of FAI if identified.

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to give informed consent for participation in the study.
* Male or Female, aged between 18 and 75 years.
* Symptomatic labral tear with evidence of labral tear on MRI.
* No radiographic evidence of OA (Kellgren-Lawrence Grade < 2)

Exclusion Criteria:

* Previous ipsilateral hip surgery
* Irreparable labral tear
* Previous fracture of femoral neck or acetabulum
* Female patient who is pregnant
* Established osteoarthritis (Kellgren-Lawrence ≥ 2)
* Hip dysplasia

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Estimated)
Dates: Start 2016-12; Primary Completion 2017-12 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Hip Outcome Score | 6 Months Post Intervention
  Change in Hip Outcome Score (Activities of Daily Living Subscale) at 6 months post intervention from baseline.

SECONDARY OUTCOMES:
Hip Outcome Scores (HOS) | 12, 18 & 24 months post intervention
  Hip Outcome Score at 12, 18 and 24 months post-operatively.
Physiologic MRI | 6 Months Post Intervention
  T2 relaxation time
X Ray | 6 Months Post Intervention
  Joint space width
X Ray | 6 Months Post Intervention
  Kellgren-Lawrence score
Biomarkers of Osteo Arthritis (OA) | At surgery and 6, 12 & 24 months post intervention.
  Biomarkers of OA from synovial fluid and serum.
Clinical Assessment of Function | 6, 12 & 24 months post intervention.
  Clinical assessment of range of motion and impingement tests.
Health Economics | 6, 12, 18 & 24 months post intervention
  Assessment of economic burden associated with disease using EQ5D score
Physiologic MRI | 6 Months Post Intervention
  T1 Rho

CONTACTS AND LOCATIONS:
Overall Officials: Sion Glyn-Jones, Principal Investigator — University of Oxford
Locations (1):
- Nuffield Orthopaedic Centre, Oxford University Hospitals Trust, Oxford, Oxfordshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No